CLINICAL TRIAL: NCT04042324
Title: A Randomized 3 Period Crossover Study to Investigate the Effect of Triferic Plus Heparin Infusion Compared to Heparin Alone on Coagulation Parameters in Hemodialysis Patients
Brief Title: A Study to Investigate the Effect of Triferic Plus Heparin Infusion Compared to Heparin Alone on Coagulation Parameters in Hemodialysis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-24
Record Dates: First submitted 2019-07-22; First posted 2019-08-01 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human); Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Triferic post-dialyzer; UFH via continuous infusion (Experimental): Patients will receive Triferic 6.75 mg IV over 3 hours into the post-dialyzer blood line (or drip chamber) administered by an infusion pump. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of heparin using the on-machine infusion pump. The infusion of heparin to be stopped at hour 3 of hemodialysis.
  Interventions: Drug: Triferic; Drug: Heparin
- UFH and Triferic admixture (Experimental): Patients will receive Triferic 6.75 mg IV plus the appropriate volume of unfractionated heparin for continuous infusion over 3 hours into the pre-dialyzer "heparin line". This mixture will be administered by the on-machine syringe infusion pump for continuous infusion. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of Triferic + heparin. The infusion of Triferic + heparin will be stopped at hour 3 of hemodialysis.
  Interventions: Drug: Triferic; Drug: Heparin
- UFH via continuous infusion pre-dialyzer (Experimental): Patients will receive no Triferic. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of heparin via the on-machine syringe pump. The infusion of heparin to be stopped at hour 3 of hemodialysis
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Triferic — Triferic (ferric pyrophosphate citrate, FPC), an iron-replacement product, is an iron complex in which iron(III) is bound to pyrophosphate and citrate.
  Other Names: ferric pyrophosphate citrate; FPC
  Arms: Triferic post-dialyzer; UFH via continuous infusion; UFH and Triferic admixture
Drug: Heparin — Unfractionated heparin (UFH): a common anticoagulant used during hemodialysis treatments.
  Other Names: Unfractionated heparin; UFH

SUMMARY:
This study will investigate the effect of co-administration of Triferic and heparin on the ability to maintain circuit anti-coagulation and iron delivery when compared to control conditions when each treatment is administered via separate routes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult hemodialysis patients ≥18 years of age.
2. Signed informed consent to participate in the study.
3. Stable on hemodialysis prescription for ≥3 months.
4. Hemoglobin concentration >9.5 g/dL.
5. Serum TSAT ≥20%.
6. Able to receive continuous heparin infusion as their anticoagulation protocol.
7. Receiving hemodialysis via AV (arteriovenous) fistula or graft.
8. Able to receive hemodialysis for 4 hours at each session over the duration of the treatment periods.

Exclusion Criteria:

1. Active bleeding disorder (GI, skin, nasal…)
2. Receiving hemodialysis via catheter.
3. Receiving heparin free dialysis.
4. Receiving low molecular weight heparin as sole anti-coagulation for dialysis.
5. Receiving IV iron within 2 weeks of the first on-study hemodialysis treatment.
6. Receiving oral anti-coagulants or anti-platelet agents.
7. Any other condition, that in the opinion of the investigator would not allow completion of the 3 hemodialysis treatments in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Pratt, MD, Study Director — Rockwell Medical
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All twelve participants enrolled in the study were randomly assigned to cross-over between the three treatments on Days 1, 3 and 5.
Groups:
- UFH and Triferic Admixture (Day 1): Patients will receive Triferic 6.75 mg IV plus the appropriate volume of unfractionated heparin for continuous infusion over 3 hours into the pre-dialyzer "heparin line". This mixture will be administered by the on-machine syringe infusion pump for continuous infusion. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of Triferic + heparin. The infusion of Triferic + heparin will be stopped at hour 3 of hemodialysis.
- Triferic Post-dialyzer; UFH Via Continuous Infusion (Day 3): Patients will receive Triferic 6.75 mg IV over 3 hours into the post-dialyzer blood line (or drip chamber) administered by an infusion pump. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of heparin using the on-machine infusion pump. The infusion of heparin to be stopped at hour 3 of hemodialysis.
- UFH Via Continuous Infusion Pre-dialyzer (Day 5): Patients will receive no Triferic. Anti-coagulation will be provided by a bolus of heparin administered into the venous return line immediately prior to the initiation of hemodialysis followed by a continuous infusion of heparin via the on-machine syringe pump. The infusion of heparin to be stopped at hour 3 of hemodialysis
Period: UFH and Triferic Admixture (Day 1)
Arm/Group | UFH and Triferic Admixture (Day 1) | Triferic Post-dialyzer; UFH Via Continuous Infusion (Day 3) | UFH Via Continuous Infusion Pre-dialyzer (Day 5)
Started | 12 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Triferic Post-dialyzer (Day 3)
Arm/Group | UFH and Triferic Admixture (Day 1) | Triferic Post-dialyzer; UFH Via Continuous Infusion (Day 3) | UFH Via Continuous Infusion Pre-dialyzer (Day 5)
Started | 0 | 12 | 0
Completed | 0 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Triferic Pre-dialyzer (Day 5)
Arm/Group | UFH and Triferic Admixture (Day 1) | Triferic Post-dialyzer; UFH Via Continuous Infusion (Day 3) | UFH Via Continuous Infusion Pre-dialyzer (Day 5)
Started | 0 | 0 | 12
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the study who received any amount of UFH, regardless of how the dose was administered.
Groups:
- Safety Population: All patients enrolled in the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Anti-Xa Activity as Measured by the AUC (Area Under the Curve) 0-t
Time Frame: 8 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | UFH and Triferic Admixture | UFH Via Continuous Infusion Pre-dialyzer
Number analyzed (Participants) | 12 | 12
IU*hr/mL | .798 (61.6) | .733 (62.4)

2. Secondary Outcome: Anti-Xa Activity as Measured by the AUC (Area Under the Curve) 0-4 Hours
Time Frame: 4 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture | UFH Via Continuous Infusion Pre-dialyzer
Number analyzed (Participants) | 12 | 12 | 12
IU*hr/mL | .581 (75.7) | .600 (77.9) | .538 (81.0)

3. Secondary Outcome: aPTT (Activated Partial Thromboplastin Time) as Measured by the AUC (Area Under the Curve) 0-4 Hours
Time Frame: 4 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture | UFH Via Continuous Infusion Pre-dialyzer
Number analyzed (Participants) | 12 | 12 | 12
IU*hr/mL | 188 (37.7) | 196 (38.5) | 188 (39.8)

4. Secondary Outcome: TT (Thrombin Time) as Measured by the AUC (Area Under the Curve) 0-4 Hours
Time Frame: 4 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture | UFH Via Continuous Infusion Pre-dialyzer
Number analyzed (Participants) | 12 | 12 | 12
IU*hr/mL | 97.6 (31.6) | 98.0 (34.6) | 104 (40.1)

5. Secondary Outcome: Iron Profile as Measured by the sFe Cmax (Peak Serum Iron Concentration)
Time Frame: 8 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/dL
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture
Number analyzed (Participants) | 12 | 12
ug/dL | 180 (20.9) | 174 (31.5)

6. Secondary Outcome: Iron Profile as Measured by the AUC (Area Under the Curve) 0-t
Time Frame: 8 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/dL
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture
Number analyzed (Participants) | 12 | 12
h*ug/dL | 1040 (31.1) | 1050 (43.4)

ADVERSE EVENTS:
Time Frame: 1.5 weeks
Description: Adverse events were collected from date of enrollment through the date of final study visit.
Arm/Group | Triferic Post-dialyzer; UFH Via Continuous Infusion | UFH and Triferic Admixture | UFH Via Continuous Infusion Pre-dialyzer
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04042324/Prot_SAP_000.pdf